CLINICAL TRIAL: NCT05818306
Title: A Phase Ia, Randomized, Parallel-group, Double-blind, Placebo-controlled, Single-center, Multiple Dose Safety and Tolerability Study of Ascending Doses of BL-001 Oral Capsules Administered for 28 Days to Healthy Volunteers
Brief Title: A Phase Ia Safety and Tolerability Study of BL-001
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Bloom Science (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Health Services Research
Other Study IDs: BL-001-1001
Record Dates: First submitted 2023-03-24; First posted 2023-04-18 (Actual); Last update posted 2023-06-27 (Actual); Status verified 2023-06

CONDITIONS: Healthy Volunteers
Keywords: Bloom Science; Bloom; BL-001; Microbiome; LBP; Live Biological Product; Live Biotherapeutic Product

STUDY DESIGN:
Intervention Model Description: Randomized, parallel-group, double-blind, placebo-controlled, single-center, multiple dose safety & tolerability Phase Ia study
Who Masked: Participant, Care Provider, Investigator
Masking Description: Both the Investigator and the subjects are not aware of the treatment administered.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (4):
- Cohort A Dose 1 (Experimental): Oral, daily administration of BL-001 Dose 1 or Placebo randomized 3:1 (BL-001: Placebo)
  Interventions: Drug: BL-001; Drug: Placebo
- Cohort B Dose 2 (Experimental): Oral, daily administration of BL-001 Dose 2 or Placebo randomized 3:1 (BL-001: Placebo)
  Interventions: Drug: BL-001; Drug: Placebo
- Cohort C Dose 3 (Experimental): Oral, daily administration of BL-001 Dose 3 or Placebo randomized 3:1 (BL-001: Placebo)
  Interventions: Drug: BL-001; Drug: Placebo
- Cohort D Dose 4 (Experimental): Oral, daily administration of BL-001 Dose 4 or Placebo randomized 3:1 (BL-001: Placebo)
  Interventions: Drug: BL-001; Drug: Placebo

INTERVENTIONS:
Drug: BL-001 — Live biological product BL-001
Drug: Placebo — Placebo

SUMMARY:
To investigate the safety and tolerability of BL-001 in healthy volunteers for 28 consecutive days.

DETAILED DESCRIPTION:
This is a Phase 1a randomized, parallel-group, double-blind, placebo-controlled, single-center, multiple dose study to evaluate the safety and tolerability of BL-001.

ELIGIBILITY:
Key Inclusion criteria

1. Informed consent: signed written informed consent before inclusion in the study
2. Sex and Age: men/women, 18-55 years old inclusive
3. Body Mass Index (BMI): 18.5-30 kg/m2 inclusive
4. Vital signs: systolic blood pressure 100-139 mmHg, diastolic blood pressure 50-89 mmHg, heart rate 50-90 bpm, measured after 5 min at rest in the sitting position
5. Full comprehension: ability to comprehend the full nature and purpose of the study, including possible risks and side effects; ability to co-operate with the investigator and to comply with the requirements of the entire study
6. Contraception and fertility (women only): women of child-bearing potential must be using at least one of the protocol defined and reliable methods of contraception

Key Exclusion criteria

1. Electrocardiogram 12-leads (supine position): clinically significant abnormalities
2. Physical findings: clinically significant abnormal physical findings which could interfere with the objectives of the study
3. Bowel movements: on average ≥3 stools per day or <3 stools per week
4. Laboratory analyses: clinically significant abnormal laboratory values indicative of physical illness
5. Allergy: ascertained or presumptive hypersensitivity to the formulation's ingredients; history of anaphylaxis to drugs or allergic reactions in general, which the Investigator considers may affect the outcome of the study
6. Diseases: significant history of renal, hepatic, gastrointestinal, cardiovascular, respiratory, skin, hematological, endocrine, psychiatric or neurological diseases that may interfere with the aim of the study
7. Gastrointestinal: evidence of acute or chronic gastrointestinal disorders
8. Medications and probiotics: probiotics, nutraceuticals, and medications, including over the counter medications and herbal remedies for 2 weeks and antibiotics for 3 months before the start of the study. Hormonal contraceptives for women will be allowed

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 32 (Actual)
Dates: Start 2023-02-20 (Actual); Primary Completion 2023-05-19 (Actual); Study Completion 2023-06-02 (Actual)

PRIMARY OUTCOMES:
Safety and tolerability of BL-001 | Treatment-emergent adverse events are reviewed from screening through Day 28
  Safety and tolerability of BL-001 as measured by treatment-emergent adverse events

SECONDARY OUTCOMES:
Intestinal engraftment | Fecal samples are collected by the subjects at home from screening through Day 28
  The intestinal engraftment of the microbiota with BL-001 component strains
Intestinal microbiota changes | Fecal samples are collected by the subjects at home from screening through Day 28
  Changes in the intestinal microbiota, including microbial taxonomic and functional characterization as well as diversity metrics
Metabolite changes in stool samples | Fecal samples are collected by the subjects at home from screening through Day 28
  Analysis of metabolite changes in stool samples
Metabolite changes in plasma samples | Venous blood samples are collected by venipuncture from a forearm vein at visits starting at screening through Day 28
  Analysis of metabolite changes in plasma samples

CONTACTS AND LOCATIONS:
Overall Officials: Paolo Baroldi, Study Director — Bloom Science
Locations (1):
- CROSS Research S.A., Arzo, Canton Ticino, Switzerland

IPD SHARING:
Plan to Share IPD: No